CLINICAL TRIAL: NCT01330381
Title: Trial Consisting of an 8-week Double-blind Placebo-controlled Part to Evaluate Efficacy, Safety, Tolerability and Pharmacokinetics of Prucalopride in Paediatric Subjects With Functional Constipation, Aged ≥6 Months to <18 Years, Followed by a 16-week Open-label Comparator (PEG) Controlled Part, to Document Safety and Tolerability up to 24 Weeks
Brief Title: Prucalopride in Pediatric Subjects With Functional Constipation
Acronym: FC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD555-303; M0001-C303 (Other: Movetis); 2010-022402-40 (EudraCT Number)
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Results first posted 2014-02-26 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Functional Constipation
MeSH Terms: interventions — prucalopride; Polyethylene Glycols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- prucalopride (Experimental): drug
  Interventions: Drug: prucalopride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PEG 4000 (Active Comparator): 4-20g administered as an oral solution once daily
  Interventions: Drug: PEG 4000

INTERVENTIONS:
Drug: prucalopride — prucalopride
  * subjects with weight ≤50kg: 0.04 mg/kg once daily as oral solution of 0.4 mg/ml
  * subjects with weight >50 kg: prucalopride 2 mg tablet once daily
  Arms: prucalopride
Drug: Placebo — Matching oral solution or oral tablets given once daily
  Arms: Placebo
Drug: PEG 4000
  Arms: PEG 4000

SUMMARY:
To evaluate the efficacy of prucalopride compared to placebo for the treatment of functional constipation in a paediatric population, aged ≥ 6 months to < 18 years. A 16-week open-label comparator (PEG) controlled part will follow, to document safety and tolerability up to 24 weeks.

ELIGIBILITY:
Main Inclusion Criteria:

1. Boys and girls, aged ≥ 6 months and < 18 years.
2. Subjects with a confirmed diagnosis of functional constipation as defined by the Rome III criteria.

Main Exclusion Criteria:

1. Children with underlying GI abnormalities and causes for defecation disorders.
2. Constipation is thought to be drug-induced.
3. Subjects suffering from secondary causes of chronic constipation.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 215 (Actual)
Dates: Start 2011-04-28 (Actual); Primary Completion 2013-03-01 (Actual); Study Completion 2013-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Academisch Medisch Centrum, Amsterdam, Netherlands

REFERENCES:
- [Result] Mugie SM, Korczowski B, Bodi P, Green A, Kerstens R, Ausma J, Ruth M, Levine A, Benninga MA. Prucalopride is no more effective than placebo for children with functional constipation. Gastroenterology. 2014 Dec;147(6):1285-95.e1. doi: 10.1053/j.gastro.2014.09.005. Epub 2014 Sep 16. PMID 25239590
- [Derived] van Schaick E, Benninga MA, Levine A, Magnusson M, Troy S. Development of a population pharmacokinetic model of prucalopride in children with functional constipation. Pharmacol Res Perspect. 2016 Jun 1;4(4):e00236. doi: 10.1002/prp2.236. eCollection 2016 Aug. PMID 27891230

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects who completed the 8 week double blind treatment period and wished to continue were re-randomized after the double-blind treatment period to the 16 week open-label treatment period. Out of 215 subjects randomized in the study, 213 subjects received treatment and 2 subjects withdrew consent before treatment.
Groups:
- Prucalopride: Subjects with weight ≤50 kg received 0.04 mg/kg prucalopride once daily as oral solution of 0.4 mg/mL. Subjects with weight >50 kg received prucalopride 2 mg oral tablet once daily.
- Placebo: Subjects with weight ≤50 kg received placebo matching to prucalopride oral solution. Subjects with weight >50 kg received placebo matching prucalopride oral tablet.
- PEG 4000 (Polyethylene Glycol): Subjects received PEG 4000 oral solution at a dose of 4 gram to 20 gram once daily.
Period: Double-blind Treatment Period (8 Weeks)
Arm/Group | Prucalopride | Placebo | PEG 4000 (Polyethylene Glycol)
Started | 107 | 108 | 0
Received Treatment | 106 | 107 | 0
Completed | 96 | 101 | 0
Not Completed | 11 | 7 | 0
Not completed — Withdrawal by Subject | 5 | 4 | 0
Not completed — Non-compliance | 2 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Did not fulfill inclusion/exclusion | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0
Period: Open-label Treatment Period (16 Weeks)
Arm/Group | Prucalopride | Placebo | PEG 4000 (Polyethylene Glycol)
Started | 98 | 0 | 99
Completed | 88 | 0 | 81
Not Completed | 10 | 0 | 18
Not completed — Withdrawal by Subject | 7 | 0 | 16
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Sponsor's decision | 1 | 0 | 1
Not completed — Non-compliance | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Set was used for baseline characteristics. The Safety Set includes all subjects who were randomized and received at least 1 dose of investigational product. One randomized subject in each group did not receive investigational product and therefore were not included in the Safety Set.
Groups:
- Placebo: Subjects with weight ≤50 kg received placebo matching to prucalopride oral solution. Subjects with weight >50 kg received placebo matching to prucalopride oral tablet.
- Total: Total of all reporting groups
Arm/Group | Prucalopride | Placebo | Total
Number analyzed (Participants) | 106 | 107 | 213
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 106 | 107 | 213
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.3 (4.54) | 8.2 (4.69) | 8.3 (4.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 58 | 118
  Male | 46 | 49 | 95
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 39 | 35 | 74
  Netherlands | 25 | 26 | 51
  Poland | 23 | 23 | 46
  United Kingdom | 10 | 10 | 20
  Belgium | 4 | 4 | 8
  Germany | 1 | 6 | 7
  France | 2 | 2 | 4
  Italy | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent of Responders in the Last Four Weeks of the Double-Blind Treatment Period
Description: Responders are defined as subjects with an average spontaneous defecation frequency is ≥3 times per week AND the average number of fecal incontinence episodes per 2 weeks is ≤ 1 episode (only for subjects after acquisition of toileting skills).
Time Frame: Last 4 weeks of double-blind treatment period
Population: Full Analysis Set includes all subjects who were randomized and received at least 1 dose of investigational product.
Measure: Number; unit: percentage of subjects
Arm/Group | Prucalopride | Placebo
Number analyzed (Participants) | 106 | 107
percentage of subjects | 17.0 | 17.8
Statistical Analysis 1: Comparison: Prucalopride vs Placebo; Test type: Superiority or Other; p = 0.9002, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percent of Subjects With Bowel Frequency of 3 or More Spontaneous Bowel Movements (SBM) Per Week in the Last Four Weeks of the Double-Blind Treatment Period
Description: Spontaneous Bowel Movements defined as a bowel movement that is not preceded within a period of 24 hours by the intake of a laxative agent or by the use of an enema.
Time Frame: Last 4 weeks of double-blind treatment period
Population: Full Analysis Set includes all subjects who were randomized and received at least 1 dose of investigational product.
Measure: Number; unit: percentage of subjects
Arm/Group | Prucalopride | Placebo
Number analyzed (Participants) | 106 | 107
percentage of subjects | 29.2 | 35.5
Statistical Analysis 1: Comparison: Prucalopride vs Placebo; Test type: Superiority or Other; p = 0.3520, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percent of Subjects With Fecal Incontinence Episodes of 1 or Less Per 2 Weeks in the Last Four Weeks of the Double-Blind Treatment Period
Description: Fecal incontinence is a lack of control over defecation, leading to involuntary loss of bowel contents (only for subjects after acquisition of toileting skills).
Time Frame: Last 4 weeks of double-blind treatment period
Population: Full Analysis Set includes all subjects who were randomized and received at least 1 dose of investigational product. Not all subjects in the Full Analysis Set had data for this outcome.
Measure: Number; unit: percentage of subjects
Arm/Group | Prucalopride | Placebo
Number analyzed (Participants) | 93 | 93
percentage of subjects | 43.0 | 43.0
Statistical Analysis 1: Comparison: Prucalopride vs Placebo; Test type: Superiority or Other; p = 0.5228, Cochran-Mantel-Haenszel

4. Secondary Outcome: Number of Retentive Posturing or Excessive Volitional Stool Retention in the Double-Blind Treatment Period
Description: Purposefully avoiding defecation.
Time Frame: Over the 8 week double blind treatment period
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: retentions/week
Arm/Group | Prucalopride | Placebo
Number analyzed (Participants) | 105 | 107
retentions/week | 1.1 (1.82) | 1.2 (1.71)

5. Secondary Outcome: Painful Bowel Movements Score in the Double-Blind Treatment Period
Description: Pain was rated on a 6-point scale (0=no hurt, 1=hurts little bit, 2=hurts little more, 3=hurts even more, 4=hurts whole lot, 5=hurts worst) in subjects of 3 years and older. Lower scores represent less pain.
Time Frame: Over the 8 week double blind treatment period
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prucalopride | Placebo
Number analyzed (Participants) | 98 | 100
units on a scale | 1.3 (1.25) | 1.7 (1.34)

6. Secondary Outcome: Stool Consistency Per SBM Score in Children Without Diapers in the Double-Blind Treatment Period
Description: Measured using the 7-point Bristol scale where 1-2 indicate constipation, 3-4 are ideal stools, and 5-7 tending toward diarrhea.
Time Frame: Over the 8 week double blind treatment period
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prucalopride | Placebo
Number analyzed (Participants) | 92 | 93
units on a scale | 3.8 (0.96) | 3.6 (1.17)

7. Secondary Outcome: Stool Consistency Per SBM Score in Children With Diapers in the Double-Blind Treatment Period
Description: Measured on a 4-point scale where 1 is constipation, 2-3 is ideal, and 4 is diarrhea.
Time Frame: Over the 8 week double blind treatment period
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prucalopride | Placebo
Number analyzed (Participants) | 13 | 14
units on a scale | 2.1 (0.47) | 2.0 (0.59)

8. Secondary Outcome: Large Diameter Stools in the Double-Blind Treatment Period
Description: Large diameter stools make defecation more difficult. Small diameter stools are better.
Time Frame: Over the 8 week double blind treatment period
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: large diameter stools/week
Arm/Group | Prucalopride | Placebo
Number analyzed (Participants) | 105 | 107
large diameter stools/week | 1.7 (1.67) | 1.7 (1.2)

9. Secondary Outcome: Abdominal Pain Score in Double-Blind Treatment Period
Description: as for outcome 5
Time Frame: Over the 8 week double blind treatment period
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prucalopride | Placebo
Number analyzed (Participants) | 96 | 95
units on a scale | 0.9 (1.18) | 1.1 (1.15)

10. Secondary Outcome: Frequency of Toilet Training in the Double-Blind Treatment Period
Description: Only for subjects after acquisition of toileting skills.
Time Frame: Over the 8 week double blind treatment period
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: toilet trainings/week
Arm/Group | Prucalopride | Placebo
Number analyzed (Participants) | 82 | 75
toilet trainings/week | 4.9 (2.47) | 5.1 (2.47)

11. Secondary Outcome: Number of Rescue Medications Taken in the Double-Blind Treatment Period
Time Frame: Over the 8 week double blind treatment period
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: rescue medications/week
Arm/Group | Prucalopride | Placebo
Number analyzed (Participants) | 105 | 107
rescue medications/week | 1.2 (1.25) | 1.3 (1.09)

12. Secondary Outcome: Time to First SBM in the Double-Blind Treatment Period
Description: After intake of the trial medication on Day 1.
Time Frame: Day 1 onwards
Population: Full Analysis Set includes all subjects who were randomized and received at least 1 dose of investigational product.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Prucalopride | Placebo
Number analyzed (Participants) | 106 | 107
hours | 67.00 [49.42 to 101.17] | 99.75 [73.75 to 204.00]
Statistical Analysis 1: Comparison: Prucalopride vs Placebo; Test type: Superiority or Other; p = 0.377, Chi-squared

13. Secondary Outcome: Number of SBM Per Week in the Double-Blind Treatment Period
Time Frame: Over the 8 week double blind treatment period
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: SBM/week
Arm/Group | Prucalopride | Placebo
Number analyzed (Participants) | 105 | 107
SBM/week | 2.3 (2.35) | 2.1 (1.74)

14. Secondary Outcome: Change From Baseline in the Number of SBM Per Week Over the 8 Week Double Blind Treatment Period
Time Frame: Baseline and over the 8 week double blind treatment period
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: SBM/week
Arm/Group | Prucalopride | Placebo
Number analyzed (Participants) | 105 | 107
SBM/week | 1.5 (2.35) | 1.0 (1.78)

15. Secondary Outcome: Severity of Constipation Over the Past 2 Weeks for the Final On Treatment Assessment in the Double-Blind Treatment Period
Time Frame: 2 weeks
Population: as for outcome 3
Measure: Number; unit: percentage of subjects
Arm/Group | Prucalopride | Placebo
Number analyzed (Participants) | 103 | 107
percentage of subjects
  Absent | 15.5 | 5.6
  Mild | 21.4 | 18.7
  Moderate | 19.4 | 27.1
  Severe | 27.2 | 24.3
  Very severe | 16.5 | 24.3
Statistical Analysis 1: Comparison: Prucalopride vs Placebo; Test type: Superiority or Other; p = 0.1599, Van Elteren test

16. Secondary Outcome: Severity of Constipation Over the Past 2 Weeks for the Final On Treatment Assessment in the Open-Label Treatment Period
Time Frame: 2 weeks
Population: as for outcome 3
Measure: Number; unit: percentage of subjects
Groups:
- PEG 4000: Subjects received PEG 4000 oral solution at a dose of 4 gram to 20 gram once daily.
Arm/Group | Prucalopride | PEG 4000
Number analyzed (Participants) | 97 | 93
percentage of subjects
  Absent | 24.7 | 46.2
  Mild | 17.5 | 16.1
  Moderate | 17.5 | 9.7
  Severe | 15.5 | 15.1
  Very severe | 24.7 | 12.9
Statistical Analysis 1: Comparison: Prucalopride vs PEG 4000; Test type: Superiority or Other; p = 0.0003, Van Elteren test

17. Secondary Outcome: Efficacy of Treatment for Final On Treatment Assessment in Double-Blind Treatment Period
Time Frame: Over the 8 week double blind treatment period
Population: as for outcome 3
Measure: Number; unit: percentage of subjects
Arm/Group | Prucalopride | Placebo
Number analyzed (Participants) | 103 | 107
percentage of subjects
  Not at all effective | 33.0 | 32.7
  Little bit effective | 14.6 | 18.7
  Moderately effective | 15.5 | 25.2
  Quite a bit effective | 22.3 | 14.0
  Extremely effective | 14.6 | 9.3
Statistical Analysis 1: Comparison: Prucalopride vs Placebo; Test type: Superiority or Other; p = 0.4647, Van Elteren test

18. Secondary Outcome: Efficacy of Treatment for Final On Treatment Assessment in Open-Label Treatment Period
Time Frame: Over the 16 week open label treatment period
Population: as for outcome 3
Measure: Number; unit: percentage of subjects
Arm/Group | Prucalopride | PEG 4000
Number analyzed (Participants) | 97 | 93
percentage of subjects
  Not at all effective | 29.9 | 15.1
  Little bit effective | 10.3 | 5.4
  Moderately effective | 20.6 | 11.8
  Quite a bit effective | 18.6 | 21.5
  Extremely effective | 20.6 | 46.2
Statistical Analysis 1: Comparison: Prucalopride vs PEG 4000; Test type: Superiority or Other; p < 0.0001, Van Elteren test

19. Secondary Outcome: Convenience of Treatment for Final On Treatment Assessment in Open-Label Treatment Period
Time Frame: Over the 16 week open label treatment period
Population: as for outcome 3
Measure: Number; unit: percentage of subjects
Arm/Group | Prucalopride | PEG 4000
Number analyzed (Participants) | 97 | 90
percentage of subjects
  Neutral | 16.5 | 15.6
  Very difficult | 1.0 | 2.2
  Quite difficult | 0.0 | 5.6
  Quite easy | 27.8 | 28.9
  Very easy | 54.6 | 47.8
Statistical Analysis 1: Comparison: Prucalopride vs PEG 4000; Test type: Superiority or Other; p = 0.3044, Van Elteren test

ADVERSE EVENTS:
Time Frame: Baseline up to Week 24
Groups:
- Prucalopride (Double-blind Period); Prucalopride (Open-label Period): Subjects with weight ≤50 kg received 0.04 mg/kg prucalopride once daily as oral solution of 0.4 mg/mL. Subjects with weight >50 kg received prucalopride 2 mg oral tablet once daily.
- Placebo (Double-blind Period): Subjects with weight ≤50 kg received placebo matching to prucalopride oral solution. Subjects with weight >50 kg received placebo matching to prucalopride oral tablet.
- PEG 4000 (Open-label Period): Subjects received PEG 4000 oral solution at a dose of 4 gram to 20 gram once daily.
Arm/Group | Prucalopride (Double-blind Period) | Placebo (Double-blind Period) | Prucalopride (Open-label Period) | PEG 4000 (Open-label Period)
Serious Adverse Events (participants affected / at risk) | 5/106 | 2/107 | 4/98 | 1/99
Other Adverse Events (participants affected / at risk) | 53/106 | 50/107 | 44/98 | 44/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prucalopride (Double-blind Period) (N=106) | Placebo (Double-blind Period) (N=107) | Prucalopride (Open-label Period) (N=98) | PEG 4000 (Open-label Period) (N=99)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prucalopride (Double-blind Period) (N=106) | Placebo (Double-blind Period) (N=107) | Prucalopride (Open-label Period) (N=98) | PEG 4000 (Open-label Period) (N=99)
Constipation (Gastrointestinal disorders) | 2 (3) | 2 (2) | 6 (8) | 2 (2)
Vomiting (Gastrointestinal disorders) | 14 (16) | 5 (5) | 9 (10) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 13 (17) | 12 (21) | 9 (9) | 11 (12)
Bronchitis (Infections and infestations) | 2 (2) | 7 (8) | 5 (5) | 3 (3)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 6 (6) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 2 (4) | 5 (7) | 5 (6) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 4 (4) | 6 (6)
Pyrexia (General disorders) | 15 (18) | 3 (4) | 5 (5) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 6 (6) | 3 (5) | 12 (13)
Headache (Nervous system disorders) | 17 (24) | 9 (11) | 3 (3) | 7 (7)
Nausea (Gastrointestinal disorders) | 9 (11) | 6 (6) | 4 (4) | 1 (1)
Viral infection (Infections and infestations) | 6 (6) | 5 (5) | 3 (4) | 4 (5)
Pharyngitis (Infections and infestations) | 3 (3) | 6 (6) | 5 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.